CLINICAL TRIAL: NCT02369848
Title: Shockwave Lithoplasty DISRUPT Trial for PAD (DISRUPT PAD 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD 0232
Record Dates: First submitted 2015-02-09; First posted 2015-02-24 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Lithoplasty Treatment (Experimental): Shockwave Lithoplasty System
  Interventions: Device: Shockwave Lithoplasty System

INTERVENTIONS:
Device: Shockwave Lithoplasty System

SUMMARY:
Shockwave Medical, Inc. intends to conduct a prospective, single-arm, multi-center, clinical study designed to evaluate the safety and performance of the Shockwave Lithoplasty™ System in subjects with moderate to heavily calcified peripheral arteries with 3.50mm to 7.0mm reference vessel diameter at the target site. The Shockwave Lithoplasty™ System is indicated to generate sonic shockwave energy within the target treatment site and disrupt calcium within the lesion to allow for subsequent dilation of a peripheral artery stenosis using low balloon pressure. Up to sixty (60) subjects will be enrolled and treated with Lithoplasty to yield thirty (51) evaluable subjects complete the study assuming a 15% lost to follow-up rate.

DETAILED DESCRIPTION:
Shockwave Medical, Inc. intends to conduct a prospective, single-arm, multi-center, clinical study designed to evaluate the safety and performance of the Shockwave Lithoplasty™ System in subjects with moderate to heavily calcified peripheral arteries with 3.50mm to 7.0mm reference vessel diameter at the target site. The Shockwave Lithoplasty™ System is indicated for lithotripsy-enhanced, low-pressure balloon dilation of calcified, stenotic peripheral arteries in patients who are candidates for percutaneous therapy. Up to sixty (60) subjects will be enrolled at up to 8 centers in Europe and New Zealand to yield at least 51 evaluable subjects (assuming a lost-to-follow up rate of 15%).

Subjects will be evaluated at discharge, 30 days, 6 months, and 12 months after enrollment/index procedure.

Primary endpoints include safety and efficacy. Safety is a composite of new-onset Major Adverse Events through 30 days. Efficacy is target lesion patency at 12 months by duplex ultrasound defined as freedom from ≥50% restenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
3. Age of subject is >18.
4. Rutherford Clinical Category 2, 3, or 4.
5. Resting ankle-brachial index (ABI) of ≤0.90, or ≤0.75 after exercise, of the target leg.
6. Estimated life expectancy >1 year.

Angiographic Inclusion Criteria:

1. Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guideline.
2. Target lesion that is located in a native de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to and ends proximal to the ostium of the anterior tibial artery).
3. Target lesion reference vessel diameter is between 3.50mm and 7.0mm by visual estimate.
4. Target zone is ≤150mm in length. Target lesion can be all or part of the 150mm zone.
5. Target lesion is ≥70% stenosis by investigator via visual estimate.
6. Subject has at least one patent tibial vessel on the target leg with runoff to the ankle (not supported by collateral circulation.) Tibial vessel patency is defined as no stenosis >50%.
7. Ability to pass the guidewire across the atherosclerotic lesion.
8. No evidence of aneurysm or acute or chronic thrombus in target vessel.
9. Calcification is at least moderate. (Presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending ≥ 50% the length of the lesion.)

Exclusion Criteria:

1. Rutherford Clinical Category 5 and 6.
2. Subject has active infection in the target leg.
3. Planned major amputation of the target leg (transmetatarsal or higher).
4. The use of chronic total occlusion (CTO) re-entry devices.
5. CTOs greater than 80 mm in length.
6. Any in-stent restenosis within the target zone.
7. Lesions within 10 mm of ostium of the SFA.
8. Highly tortuous arteries (bends greater than 30 degrees over the arc length of the balloon).
9. Target lesion within native or synthetic vessel grafts.
10. History of prior endovascular or surgical procedure on the index limb within the past 30 days.
11. Subject has significant stenosis (>50% stenosis) or occlusion of inflow tract before target treatment zone (e.g. iliac or common femoral) not successfully treated with Plain old Balloon Angioplasty (POBA) or stent and without complications.
12. Subject requires treatment of a peripheral lesion on the ipsilateral limb distal and beyond the 150mm target zone at the time of the enrollment/index procedure.
13. Subject has a known coagulopathy or has a bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter, or International Normalized Ratio (INR) >1.5.
14. Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated.
15. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
16. Subject has known allergy to urethane, nylon, or silicone.
17. Myocardial infarction within 60 days prior to enrollment.
18. History of stroke within 60 days prior to enrollment.
19. History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to enrollment.
20. History of thrombolytic therapy within two weeks of enrollment.
21. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L), or on dialysis.
22. Subject is pregnant or nursing.
23. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
24. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Universitäts-Herzzentrum Freiburg & Bad Krozingen
Locations (8):
- Austria (3):
  - Universitätsklinikum LKH Graz, Graz
  - Hanusch Krankenhaus, Vienna
  - Medizinische Universitat Wien, Vienna
- Germany (4):
  - Universitäts-Herzzentrum Freiburg & Bad Krozingen, Bad Krozingen
  - University Leipzig Medical Centre, Leipzig
  - St. Franziskus Hospital, Münster
  - RoMed Klinikum Rosenheim, Rosenheim
- Auckland City Hospital, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment and enrollment took place at eight clinical sites in Austria, Germany and New Zealand between August 2015 and December 2015. A total of 60 subjects with calcified, stenotic peripheral arteries were enrolled and treated with the device.
Groups:
- Shockwave Medical Inc. Peripheral Lithoplasty: The Shockwave Medical Inc. Peripheral Lithoplasty System is a proprietary lithotripsy-enhanced balloon catheter system designed to be delivered through the peripheral arterial system of the lower extremities to the site of a calcified stenosis. Activating the lithotripsy within the device will generate pulsatile mechanical energy within the target treatment site, disrupt calcium within the lesion and allow subsequent dilation of a peripheral artery stenosis using low balloon pressure. The system consists of a balloon catheter with multiple integrated lithotripsy emitters and generator.
Period: Overall Study
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Started | 60
30 Day Primary Safety Endpoint | 58
12 Month Primary Endpoint | 30
Completed | 56
Not Completed | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 60
Number analyzed (participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 57
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 6
  Austria | 30
  Germany | 24

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness Endpoint Defined as Number of Participants withTarget Lesion Patency by Duplex Ultrasound Defined as Freedom From ≥50% Restenosis
Time Frame: 12 months post-procedure
Population: Data reflects number for participants who have an evaluable (diagnostic) scheduled or unscheduled duplex ultrasound based on reporting windows and slotting rules in the Statistical Plan. Thirty out of 43 participants achieved target lesion patency.
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 43
Participants | 30

2. Primary Outcome: Safety Endpoint Defined as Composite of New-onset Major Adverse Events (MAEs)
Description: Need for emergency surgical revascularization of target limb. Unplanned target limb amputation (above the ankle). Symptomatic thrombus or distal emboli, defined as clinical signs or symptoms of thrombus or distal emboli detected in the treated limb in the area of the treated lesion or distal to the treated lesion after the index procedure and results in extended hospitalization or noted angiographically, and requiring mechanical or pharmacologic means to improve flow and results in extended hospitalization.
  Perforations and dissections of grade D or greater that require an intervention to resolve, including bail-out stenting.
Time Frame: Within 30 days following procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 59
Participants | 58

3. Secondary Outcome: Safety Measured by Number of Participants With Freedom From Major Adverse Events (MAEs)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 57
Participants | 56

4. Secondary Outcome: Secondary Endpoint of Acute Procedural Success Achieved in Number of Participants
Description: 1. The ability of the Shockwave Lithoplasty System to achieve a post-Shockwave residual diameter stenosis of <50% (with or without adjunctive Percutaneous Transluminal Angioplasty (PTA) therapy) as assessed by quantitative angiography via core lab evaluation.
  2. The ability of the Shockwave Lithoplasty System to achieve a post-Shockwave residual diameter stenosis of <50% (without adjunctive PTA therapy) as assessed by quantitative angiography via core lab evaluation.
Time Frame: Day of Procedure
Population: Full Analysis Cohort - All subjects who were enrolled in the study and where delivery of the Shockwave Medical Peripheral Lithoplasty treatment was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 60
Participants | 58

5. Secondary Outcome: Secondary Patency Measured by Number of Participants With Target Lesion Patency by Duplex Ultrasound Defined as Freedom From ≥50% Restenosis.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 43
Participants | 30

6. Secondary Outcome: Secondary Patency Measured by Number of Participants With Target Lesion Patency (Without Adjunctive PTA) by Duplex Ultrasound Defined as Freedom From ≥50% Restenosis.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 42
Participants | 30

7. Secondary Outcome: Clinical Success - Improvement of Ankle-Brachial Index (ABI) of the Target Limb.
Description: The ankle-brachial pressure index or ankle-brachial index is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm. It has been shown to be a specific and sensitive metric for the diagnosis of Peripheral Arterial Disease (PAD).
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Percent change in ABI from baseline
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 55
Percent change in ABI from baseline | 0.3 [0.2 to 0.3]

8. Secondary Outcome: Clinical Success - Improvement of Ankle-Brachial (ABI) of the Target Limb.
Description: as for outcome 7
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percent change in ABI from baseline
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 53
Percent change in ABI from baseline | 0.2 [0.2 to 0.3]

9. Secondary Outcome: Clinical Success
Description: Change in Rutherford Clinical Category at from Baseline to 6 months.
  There are seven stages to consider:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: change in Rutherford score from baseline
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 58
change in Rutherford score from baseline | -2.0 [-2.31 to -1.76]

10. Secondary Outcome: Clinical Success
Description: Change in Rutherford Clinical Category from Baseline to12 months.
  There are seven stages to condsider:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: change in Rutherford score from baseline
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 56
change in Rutherford score from baseline | -2.1 [-2.33 to -1.78]

11. Secondary Outcome: Clinical Success
Description: Change in Rutherford Clinical Category from Baseline to 30 days
  There are seven stages to condsider:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: change in Rutherford score from baseline
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
Number analyzed (Participants) | 58
change in Rutherford score from baseline | -2.3 [-2.52 to -2.10]

ADVERSE EVENTS:
Time Frame: through 30 days, 6 months, 12 months
Arm/Group | Shockwave Medical Inc. Peripheral Lithoplasty
All-Cause Mortality (participants affected / at risk) | 1/60
Serious Adverse Events (participants affected / at risk) | 31/60
Other Adverse Events (participants affected / at risk) | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shockwave Medical Inc. Peripheral Lithoplasty (N=60)
Anaemia Of Malignant Disease (Blood and lymphatic system disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Heart Valve Incompetence (Cardiac disorders) | 1 (1)
Tricuspid Valve Incompetence (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 6 (6)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioplasty (Surgical and medical procedures) | 3 (3)
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 1 (1)
Stent Placement (Surgical and medical procedures) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3 (3)
Peripheral Artery Stenosis (Vascular disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shockwave Medical Inc. Peripheral Lithoplasty (N=60)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 4 (4)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Eczema Infected (Infections and infestations) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Skin Bacterial Infection (Infections and infestations) | 1 (1)
Tinea Pedis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 15 (15)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Bleeding Varicose Vein (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Peripheral Embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No